CLINICAL TRIAL: NCT05554029
Title: Coronaphobia in Rheumatic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Collaborators: Firat University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Assistant professor, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-23
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Rheumatic Diseases
Keywords: coronaphobia; Rheumatic diseases; COVID-19
MeSH Terms: conditions — Rheumatic Diseases; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients with rheumatic diseases
  Interventions: Diagnostic Test: Coronaphobia

INTERVENTIONS:
Diagnostic Test: Coronaphobia — Coronophobia will be assessed with COVID-19-phobia scale.

SUMMARY:
COVID-19 is a contagious respiratory disease that is caused Severe Acute Respiratory Syndrome causing Coronavirus-2 (SARS-CoV-2). The most common symptoms are fever, cough and dyspnoea. Patients with rheumatic diseases are at higher risk of infections because of disease activity and immunosuppression. In addition, old age and having concomitant chronic disease are among risk factors for coronavirus. Therefore, national health services recommend patients to practice self-isolation and self-quarantine.

DETAILED DESCRIPTION:
COVID-19 is a contagious respiratory disease that is caused Severe Acute Respiratory Syndrome causing Coronavirus-2 (SARS-CoV-2). It was firstly seen in December 2019 in Wuhan, China and spread rapidly all over the world. World Health Organization (WHO) was declared COVID-19 as a pandemic in March 2020. The most common symptoms are fever, cough and dyspnoea. Social isolation and staying home have been suggested to reduce the spreading rate of COVID-19 pandemic in many countries. In addition, curfew except necessity was applied in some countries and time of curfew varied by country. Therefore, pandemic caused changes in routine life for millions of people. Patients with rheumatic diseases are at higher risk of infections because of disease activity and immunosuppression. In addition, old age and having concomitant chronic disease are among risk factors for coronavirus. Therefore, national health services recommend patients to practice self-isolation and self-quarantine. However, social isolation was concluded with more increased physical inactivity and sedentary lifestyle. The aim of this study is to investigate coronaphobia in rheumatic diseases and compare with healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 65
* Have diagnosed with Romatoid Arthritis, Ankylosing Spondylitis, Systemic Lupus Erthematosus or Fibromyalgia

Exclusion Criteria:

* Being pregnant
* Diagnosed with malignancy
* Had changes of medical treatment in the last 3 months
* Had dysfunction that limited physical activity such as severe neurological impairment, immobility or cooperation deficits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Covid-19 Phobia Scale | 2 minutes
  Covid-19 Phobia Scale (C19P-S) was developed by Arpaci et al. C19P-S is a self-reported questionnaire consisting of 20 items and four, i.e., psychological, psychosomatic, economic, and social, subscales. All items are rated on a 5-point scale from "strongly disagree" to "strongly agree". The total score ranges from 20 to 100 points;,the higher the score, the higher is the level of coronaphobia.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 3 minutes
  It consists of 14 questions that which 7 of them evaluate depression and 7 of them evaluate anxiety. Each question is scored from 0 to 3 and high scores indicate severe anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Songul B Yentur, Principal Investigator — Gazi University
Locations (1):
- Songul Baglan Yentur, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No